CLINICAL TRIAL: NCT07038954
Title: Evaluation of Stone Composition in Patients With Kidney Stones Undergoing Surgical Intervention at Binh Dan Hospita
Brief Title: Evaluation of Stone Composition in Surgical Kidney Stone Patients in Vietnam
Acronym: STONE-VN
Status: Completed | Type: Observational
Sponsor: Binh Dan Hospital (Other)
Collaborators: Department of Science and Technology of Ho Chi Minh City (Unknown)
Responsible Party: Sponsor
Other Study IDs: BDH-STONE-2023; 22441 (Other: University of Medicine and Pharmacy at Ho Chi Minh City (UMP HCMC))
Record Dates: First submitted 2025-06-05; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Kidney Stones; Urolithiasis; Nephrolithiasis
Keywords: Kidney stone composition; Percutaneous nephrolithotomy; Stone analysis; Infrared spectroscopy; Calcium oxalate; Vietnam; Binh Dan Hospital; Surgical stone treatment; Recurrent kidney stones
MeSH Terms: conditions — Kidney Calculi; Urolithiasis; Nephrolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Kidney stone fragments collected during surgical procedures, including percutaneous nephrolithotomy (PCNL), ureteroscopic lithotripsy, laparoscopic ureterolithotomy, and open stone removal. Samples were retained for compositional analysis using X-ray diffraction (XRD) and infrared spectroscopy (IR). No blood, tissue, or DNA-based samples were collected or retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgically Treated Kidney Stone Patients: This cohort includes patients aged 15 years and older who underwent surgical treatment for kidney or ureteral stones at Binh Dan Hospital between July and December 2023. Surgical methods included percutaneous nephrolithotomy (PCNL), semirigid ureteroscopic lithotripsy, laparoscopic ureterolithotomy, and open surgery. Retrieved stone fragments were analyzed using X-ray diffraction (XRD) and infrared spectroscopy (IR) to determine stone composition. No experimental intervention was applied.
  Interventions: Other: Stone Composition Analysis

INTERVENTIONS:
Other: Stone Composition Analysis — This intervention involves the compositional analysis of kidney stone fragments retrieved during surgical procedures. The stone samples are analyzed using X-ray diffraction (XRD) and infrared spectroscopy (IR) to determine their crystal composition. This is a non-invasive, laboratory-based diagnostic procedure. No drug, device, or therapeutic intervention was administered to participants as part of this observational study.

SUMMARY:
This is a prospective observational study conducted at Binh Dan Hospital, Ho Chi Minh City, Vietnam, from July to December 2023. The study aims to analyze the composition of kidney stones in patients undergoing surgical interventions such as percutaneous nephrolithotomy (PCNL), ureteroscopic lithotripsy, laparoscopic ureterolithotomy, or open surgery. Stone fragments collected during the procedures were analyzed using X-ray diffraction (XRD) and infrared spectroscopy (IR).

The primary goal of this study is to identify the types and distribution of kidney stone compositions in a Vietnamese surgical cohort and compare them with global patterns. Findings from this study are expected to provide insights into age- and gender-related differences in stone composition, and contribute to improved prevention strategies for recurrent urolithiasis.

The study was approved by the Ethics Committee of the University of Medicine and Pharmacy at Ho Chi Minh City. All participants provided written informed consent.

DETAILED DESCRIPTION:
Kidney stone disease (urolithiasis) is a common and recurrent condition worldwide. Vietnam is located in a high-incidence zone known as the "stone belt." Understanding the composition of kidney stones is essential for guiding treatment decisions and implementing effective preventive strategies. Although surgical treatment options have advanced, stone recurrence remains a significant concern. However, there is currently limited data in Vietnam regarding the composition of stones in patients undergoing surgical management.

This prospective observational study is being conducted at the Department of Urology, Binh Dan Hospital, Ho Chi Minh City, Vietnam. The study period is from July to December 2023. Eligible participants include patients aged 15 years and older undergoing surgical stone removal via one of the following procedures: percutaneous nephrolithotomy (PCNL), semirigid ureteroscopic lithotripsy, laparoscopic ureterolithotomy, or open surgery. Patients with missing or unsuitable stone samples, incomplete clinical data, or contraindications to surgery are excluded.

During surgery, retrieved stone fragments are collected for analysis. Stone composition is analyzed using both X-ray diffraction (XRD) and infrared spectroscopy (IR), which are reliable methods for identifying stone components. The analysis focuses on determining the presence of calcium oxalate (monohydrate and dihydrate), phosphate (hydroxyapatite and brushite), uric acid, infection-related stones (struvite and ammonium hydrogen urate), and cystine stones.

This study has received ethical approval from the Ethics Committee of the University of Medicine and Pharmacy at Ho Chi Minh City (Approval No. 22441-DHYD). All participants provide written informed consent prior to enrollment. The study is funded by the Department of Science and Technology of Ho Chi Minh City as part of a provincial-level research initiative, with additional institutional support from Binh Dan Hospital and the University of Medicine and Pharmacy at Ho Chi Minh City.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15 years and older.
* Diagnosed with kidney or ureteral stones requiring surgical intervention.
* Underwent PCNL, URS, laparoscopic ureterolithotomy, or open stone surgery.
* Provided written informed consent.

Exclusion Criteria:

* Patients with missing or unsuitable stone samples.
* Patients with incomplete clinical data.
* Patients with contraindications to surgery.
* Pregnant women

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with kidney stones who underwent surgical treatment at Binh Dan Hospital from July to December 2023 and consented to stone analysis.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of stone types in surgically treated kidney stone patients | Within 1 month after surgical stone removal
  Determination of the proportion of each major stone type (calcium oxalate, phosphate, uric acid, struvite, and cystine) using X-ray diffraction (XRD) and infrared spectroscopy (IR).

CONTACTS AND LOCATIONS:
Locations (1):
- Binh Dan Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-center observational study with no plan for external data requests. The dataset contains identifiable clinical and imaging information, and there is no established data-sharing protocol for this study.